CLINICAL TRIAL: NCT05816096
Title: Atraumatic Restoration Treatment Compared to the Hall Technique for Management Hypomineralization Second Primary Molars
Brief Title: ART Compared to the Hall Technique for Management HSPM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Restoration for HSPM
Record Dates: First submitted 2023-03-28; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Hypomineralization, Tooth
Keywords: ART; Hall technique; HSPM; Children; Restoration
MeSH Terms: conditions — Dental Enamel Hypomineralization

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, crossover clinical study, comparison of ART and Hall Technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Hall Technique) (Active Comparator): 31 child will be treated by one performed metal crown using Hall technique on one of HSPM affected tooth.
  The correct size of SSC for tooth will be selected. Use the separating rubber if necessary. Dried the tooth and cemented the SSC by glass ionomer luting cement and used finger pressure to seat the crown and instructed the child to bite down on the SSC.
  Half of the total number of children will received performed metal crown at the first by divided them randomly to the two groups using the randomization table.
  Interventions: Combination Product: Hall technique
- B (ART) (Experimental): 31 child will be treated by Bulk fill glass hybrid restorative system (Equia Forte HT®) using Atraumatic restoration treatment on one of HSPM affected tooth.
  Isolate the tooth by cotton rolls, remove the carious soft tissue using hand instrument excavators then condition the cavity with a polyacrylic acid solution 11.5% for 10 seconds. After washed and dried the cavity insert the GIC and protect it by Equia forte coat.
  Half of the total number of children will received ART at the first by divided them randomly to the two groups using the randomization table.
  Interventions: Combination Product: ART

INTERVENTIONS:
Combination Product: Hall technique — The child will be placed to them SSC on one of their HSPM affected teeth. Pain during treatment will be assessed using the FLACC scale and satisfaction the child and parent will be evaluated using likert scale after the treatment immediately and after one month and evaluate the success restoration adapted from Innes et al. after 3_6_9_12 month.
  Other Names: A
  Arms: A (Hall Technique)
Combination Product: ART — The child will be restored to them one of their HSPM affected teeth by GIC. Pain during treatment will be assessed using the FLACC scale and satisfaction the child and parent will be evaluated using likert scale after the treatment immediately and after one month and evaluate the success restoration adapted from Innes et al. after 3_6_9_12 month.
  Other Names: B
  Arms: B (ART)

SUMMARY:
Aims: Evaluation of treatment success on HSPM-affected molars after ART and Hall technique.

comparison of pain during treatment with ART and Hall technique in HSPM. comparison of child and parent satisfaction with restorations used by ART and Hall technique.

Design: A randomized, controlled, crossover clinical study including thirty children.

DETAILED DESCRIPTION:
Background and Aims:

Despite the widespread prevalence of HSPM:

there are no comparative studies yet between ART and Hall technique in the restoration of HSPM.

there are no studies yet on the success of ART in the treatment of HSPM.

Design:

A randomized, controlled, crossover clinical study including thirty children Each child will apply both of ART and Hall technique to him.

ELIGIBILITY:
Inclusion Criteria:

* Absolute positive, positive or negative behavior according to the Frankel Scale.
* Healthy, both physically and mentally.
* Do not take medications that interfere with the assessment of pain within 24 hours prior to treatment.
* A child with HSPM-affected primary second molars on the right and left side in one jaw.
* The HSPM affected teeth from 2-6 degree in Ghanim scale.
* Teeth with atypical carious lesions.
* Teeth with post-eruption destroyed
* The presence of a clear, intact dentinal bridge between the caries and pulp radially.

Exclusion Criteria:

* Allergy to the substances used in restoration.
* Presence of general or developmental medical conditions.
* Teeth with pulpitis inflammation or apical lesion or non-restorable.
* Teeth closed to being replaced.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Estimated)
Dates: Start 2023-03-26 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Dental pain assessed by FLACC scale | During the placement of the restoration
  Evaluated by outcome assessor using the faces, legs, activity, cry, consolability behavioral rating scale (FLACC scale) a behavioral pain assessment scale which has five criteria face, legs, activity, cry, consolability, which are each assigned a score of 0,1 or2.
  Total score of scale is summed in range 0 to10, where:0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain.

SECONDARY OUTCOMES:
Child Satisfaction with the restoration assessed by the Likert scale | Immediately after the placement of the restoration
  Self-assessment by the children using Likert scale which is a psychometric scale has five responses (very satisfied, satisfied, neutral, unsatisfied, very unsatisfied)
Parent Satisfaction with the restoration assessed by the Likert scale | Immediately after the placement of the restoration after asking the child
  Self-assessment by the parent using Likert scale which is a psychometric scale has five responses (very satisfied, satisfied, neutral, unsatisfied, very unsatisfied)
Child Satisfaction with the restoration assessed by the Likert scale | After one month from treatment
  Self-assessment by the children using Likert scale which is a psychometric scale has five responses (very satisfied, satisfied, neutral, unsatisfied, very unsatisfied)
Parent Satisfaction with the restoration assessed by the Likert scale | After one month from treatment after asking the child
  Self-assessment by the parent using Likert scale which is a psychometric scale has a five responses (very satisfied, satisfied, neutral, unsatisfied, very unsatisfied)

OTHER OUTCOMES:
Clinical success of restoration assessed by evaluation criteria for restoration assessments after 3 months | After 3 months from treatment
  Evaluated by outcome assessor using evaluation criteria for restoration assessments which has three scores (success, minor failures, major failures) for ART and Hall technique.
Radiological success of restoration assessed by Radiological success cireteria after 6 months | After 6 months from traetment
  Evaluated by outcome assessor using Radiological success cireteria for restoration.
  where the case is considered successful radiologically when all signs of pulpal necrosis are absent.
Clinical success of restoration assessed by evaluation criteria for restoration assessments after 6 months | After 6 months from treatment
  Evaluated by outcome assessor using evaluation criteria for restoration assessments which has three scores (success, minor failures, major failures) for ART and Hall technique.
Clinical success of restoration assessed by evaluation criteria for restoration assessments after 9 months | After 9 months from treatment
  Evaluated by outcome assessor using evaluation criteria for restoration assessments which has three scores (success, minor failures, major failures) for ART and Hall technique.
Clinical success of restoration assessed by evaluation criteria for restoration assessments after 12 months | After 12 months from treatment
  Evaluated by outcome assessor using evaluation criteria for restoration assessments which has three scores (success, minor failures, major failures) for ART and Hall technique.
Radiological success of restoration assessed by Radiological success cireteria after 12 months | After 12 months from treatment
  Evaluated by outcome assessor using Radiological success cireteria for restoration.
  where the case is considered successful radiologically when all signs of pulpal necrosis are absent.

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Raslan, Dr, Study Chair — Tishreen University; Aya Adl, Dr, Principal Investigator — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Undecided
Up to date, there is no decision about IPD sharing